CLINICAL TRIAL: NCT02719561
Title: Fatigue Intervention Co-design Study in Teenagers and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Spathis (Other)
Responsible Party: Sponsor-Investigator, Anna Spathis, Consultant in Palliative Medicine, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A093987
Record Dates: First submitted 2016-03-17; First posted 2016-03-25 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fatigue intervention (Experimental): Fatigue Intervention is to be co-designed by participants, and likely to include education, energy conservation and activity promotion. Participants will also decide the name of the Fatigue Intervention
  Interventions: Behavioral: Fatigue Intervention

INTERVENTIONS:
Behavioral: Fatigue Intervention — The Fatigue Intervention will include education, energy conservation and activity promotion

SUMMARY:
Fatigue is one of the most common and distressing symptoms in teenage and young adult cancer patients. Despite this, there has been virtually no research evaluating treatment for cancer-related fatigue in this young patient group. The investigators are undertaking a small qualitative study to co-design a fatigue intervention, that will then be evaluated in future research to assess its effectiveness.

DETAILED DESCRIPTION:
This small qualitative study will involve 7-10 patients who are within one year of completing cancer treatment, as well as some parents. Participants will be recruited from one centre, the Cambridge Teenage and Young Adult cancer Principal Treatment Centre. The three phases will involve a) participants being interviewed individually and attending a focus group, b) patients receiving the prototype co-designed intervention, and c) participants being interviewed after the intervention to provide feedback to allow further refinement of the intervention. The intervention will be delivered by an Allied Health Professional in the setting that participants have chosen. It is likely to involve, at a minimum, education about fatigue and support with increasing activity. It will not include administration of any medication.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Aged 16-27 with a diagnosis of cancer
* Currently or previously known to the Cambridge Teenage and Young Adult cancer service
* Primary cancer treatment completed within one year of recruitment OR on maintenance treatment for leukaemia.
* A screening score of ≥5 in a 10-item numerical rating scale of fatigue severity over the last month
* Able to give informed consent

Parents:

* The parent of a patient participant or a patient who would be eligible to participate
* The patient consents to the parent being approached about the study
* The parent is able to give informed consent

Exclusion Criteria:

* Current participation in another clinical trial

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Participant-reported feedback on design content as assessed via interviews | 3 months
Participant-reported feedback on design acceptability as assessed via interviews | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spathis, MA MB BChir, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No